CLINICAL TRIAL: NCT02451358
Title: Immunogenicity and Safety of a Single Dose or Two Doses Given 28 Days Apart of a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route in Subjects Aged 6 Months or Older in India
Brief Title: Study of a Single Dose or Two Doses of a Quadrivalent Influenza Vaccine in Subjects Aged 6 Months or Older in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QIV06; U1111-1143-8370 (Other: WHO); CTRI/2015/05/005770 (Other: CTR-India)
Record Dates: First submitted 2015-05-14; First posted 2015-05-22 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent Inactivated Influenza Vaccine (QIV)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months (Experimental): Participants aged 6 to 35 months received 2 doses of 0.25 mL QIV (2016-2017 NH formulation) intramuscularly, 1 injection each at Day 0 and 28.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine (2016-2017 NH formulation), No Preservative
- Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years (Experimental): Participants aged 3 to 8 years received 2 doses of 0.5 mL QIV (2016 SH formulation) intramuscularly, 1 injection each at Day 0 and 28.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine (2016 SH formulation), No Preservative
- Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years (Experimental): Participants aged 9 to 17 years received 1 dose of 0.5 mL QIV (2015-2016 NH formulation) intramuscularly, at Day 0.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine (2015-2016 NH formulation), No Preservative
- Quadrivalent Influenza Vaccine Group 4: >=18 Years (Experimental): Participants aged >=18 years received 1 dose of 0.5 mL QIV (2015 SH formulation) intramuscularly, at Day 0.
  Interventions: Biological: Quadrivalent Inactivated Influenza Vaccine (2015 SH formulation), No Preservative

INTERVENTIONS:
Biological: Quadrivalent Inactivated Influenza Vaccine (2016-2017 NH formulation), No Preservative — 0.25 mL, Intramuscular
  Other Names: QIV, No Preservative
  Arms: Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months
Biological: Quadrivalent Inactivated Influenza Vaccine (2016 SH formulation), No Preservative — 0.5 mL, Intramuscular
  Other Names: QIV, No Preservative
  Arms: Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years
Biological: Quadrivalent Inactivated Influenza Vaccine (2015-2016 NH formulation), No Preservative — 0.5 mL, Intramuscular
  Other Names: QIV, No Preservative
  Arms: Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years
Biological: Quadrivalent Inactivated Influenza Vaccine (2015 SH formulation), No Preservative — 0.5 mL, Intramuscular
  Other Names: QIV, No Preservative
  Arms: Quadrivalent Influenza Vaccine Group 4: >=18 Years

SUMMARY:
The aim of the study was to generate immunogenicity and safety data in the whole population to support registration of the Quadrivalent Influenza Vaccine (QIV) in India:

Primary objective:

* To describe in each age group the immune response induced by a single injection (participants aged >9 years) or 2 injections (participants aged 6 months to 8 years) of QIV.

Secondary objective:

* To describe in each age group the safety profile of QIV.

DETAILED DESCRIPTION:
All participants were vaccinated with the QIV (split-virion, inactivated) Northern Hemisphere (NH) or Southern Hemisphere (SH) formulations by the intramuscular (IM) route. Immunogenicity of the vaccine was assessed at baseline (Day 0) and 28 days after the last injection. Safety data were collected up to 28 days after each injection. Serious adverse events (SAEs) were collected throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months or older on the day of inclusion
* For participants aged 6 to 35 months only: born at full term of pregnancy (>=37 weeks) or birth weight >=2.5 kg or both
* Informed consent form had been signed and dated by the participants / participants' parent(s) or another legally acceptable representative and by an independent witness, if required by local regulations. For participants aged 7 to 17 years of age, assent form has been signed and dated by the participants
* Participants / participants' parent/legally acceptable representative were able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* For participants aged 9 years or older only: participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following any trial vaccination (except Oral Poliomyelitis Vaccine (OPV) received during national immunization days)
* For participants aged 9 years or older only: previous vaccination against influenza (in the previous 9 months) with any influenza vaccine
* For participants aged 6 months to 8 years only: previous priming with any influenza vaccine (i.e., participants who received 2 doses for at least 1 previous influenza season)
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported history of seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C, after questioning
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia or as reported by the parent/legally acceptable representative, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* For participants aged 9 years or older only: current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (axillary temperature >=38.0 degree Celsius). A prospective participants should not be included in the study until the condition had resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-07-27; Primary Completion 2017-01-28 (Actual); Study Completion 2017-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (8):
- India (8):
  - Vadodara, Gujarat
  - Mandya, Karnataka
  - Pune, Maharashtra
  - Mumbai, Parel
  - Pimpri, Pune
  - Ludhiana, Punjab
  - Kolkata, West Bengal
  - Bangalore

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 8 centers in India from 27 July 2015 to 26 November 2016.
Pre-assignment Details: A total of 400 participants (100 in each group) were enrolled and vaccinated in the study.
Groups:
- Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months: Participants aged 6 to 35 months received 2 doses of 0.25 mL Quadrivalent Influenza Vaccine (QIV) (2016-2017 Northern Hemisphere (NH) formulation) intramuscularly, 1 injection each at Day 0 and 28.
- Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years: Participants aged 3 to 8 years received 2 doses of 0.5 mL QIV (2016 Southern Hemisphere (SH) formulation) intramuscularly, 1 injection each at Day 0 and 28.
Period: Overall Study
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years
Started | 100 | 100 | 100 | 100
Vaccinated at Day 0 | 100 | 100 | 100 | 100
Vaccinated at Day 28 | 99 | 98 | 0 (Participants aged 9 years and older received only 1 dose of Quadrivalent Influenza Vaccine.) | 0 (Participants aged 9 years and older received only 1 dose of Quadrivalent Influenza Vaccine.)
Completed | 99 | 98 | 99 | 100
Not Completed | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed using Full Analysis Set (FAS) which included all participants who received at least 1 dose of vaccine and had at least 1 valid post-vaccination serology result.
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years | Total
Number analyzed (Participants) | 99 | 98 | 99 | 100 | 396
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.0 (0.8) | 4.9 (1.5) | 11.7 (2.2) | 48.5 (18.8) | 16.6 (21.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 60 | 50 | 34 | 189
  Male | 54 | 38 | 49 | 66 | 207
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 99 | 98 | 99 | 100 | 396

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies
Description: Anti-influenza antibodies were measured using hemagglutination inhibition (HAI) assay for 4 strains: H1N1, H3N2, B Victoria, B Yamagata.
Time Frame: Day 0 (pre-vaccination) and 28 days post-final vaccination (post-vaccination)
Population: Analysis was performed using Full Analysis Set (FAS) which included all participants who received at least 1 dose of vaccine and had at least 1 valid post-vaccination serology result. Here, 'Number Analyzed' = those participants with available data for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years
Number analyzed (Participants) | 99 | 98 | 99 | 100
Titers (1/dilutions)
  Pre-Vaccination: A/H1N1: number analyzed (Participants) | 99 | 98 | 99 | 99
  Pre-Vaccination: A/H1N1 | 14.4 [9.83 to 21.1] | 84.1 [53.6 to 132] | 107 [83.4 to 138] | 44.3 [31.8 to 61.6]
  Pre-Vaccination: A/H3N2 | 44.4 [26.6 to 74.2] | 416 [311 to 555] | 204 [150 to 277] | 20.8 [15.8 to 27.3]
  Pre-Vaccination: B Victoria: number analyzed (Participants) | 99 | 97 | 99 | 98
  Pre-Vaccination: B Victoria | 21.5 [14.0 to 32.8] | 37.5 [23.8 to 59.1] | 54.1 [41.4 to 70.6] | 41.9 [31.9 to 55.0]
  Pre-Vaccination: B Yamagata: number analyzed (Participants) | 99 | 98 | 99 | 99
  Pre-Vaccination: B Yamagata | 12.0 [8.82 to 16.3] | 81.1 [53.9 to 122] | 91.7 [67.2 to 125] | 107 [79.5 to 144]
  Post-Vaccination: A/H1N1: number analyzed (Participants) | 99 | 98 | 99 | 99
  Post-Vaccination: A/H1N1 | 723 [527 to 993] | 1895 [1550 to 2318] | 1641 [1398 to 1927] | 1232 [969 to 1565]
  Post-Vaccination: A/H3N2 | 1016 [697 to 1482] | 3458 [3011 to 3971] | 2379 [1994 to 2838] | 980 [736 to 1306]
  Post-Vaccination: B Victoria | 658 [441 to 982] | 2222 [1820 to 2713] | 2061 [1622 to 2617] | 1150 [913 to 1447]
  Post-Vaccination: B Yamagata: number analyzed (Participants) | 99 | 98 | 99 | 98
  Post-Vaccination: B Yamagata | 951 [675 to 1338] | 3582 [3054 to 4201] | 2273 [1750 to 2951] | 1836 [1413 to 2385]

2. Primary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: H1N1, H3N2, B Victoria and B Yamagata. Seroprotection was defined as an antibody titer >=40 (1/dilution[dil]) at pre-vaccination and at post-final vaccination.
Time Frame: Day 0 (pre-vaccination) and 28 days post-final vaccination (post-vaccination)
Population: Analysis was performed using FAS which included all participants who received at least 1 dose of vaccine and had at least 1 valid post-vaccination serology result. Here, 'Number Analyzed' = those participants with available data for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years
Number analyzed (Participants) | 99 | 98 | 99 | 100
Participants
  Pre-Vaccination: A/H1N1: number analyzed (Participants) | 99 | 98 | 99 | 99
  Pre-Vaccination: A/H1N1 | 23 | 62 | 86 | 60
  Pre-Vaccination: A/H3N2 | 40 | 94 | 85 | 34
  Pre-Vaccination: B Victoria: number analyzed (Participants) | 99 | 97 | 99 | 98
  Pre-Vaccination: B Victoria | 30 | 47 | 63 | 53
  Pre-Vaccination: B Yamagata: number analyzed (Participants) | 99 | 98 | 99 | 99
  Pre-Vaccination: B Yamagata | 18 | 65 | 74 | 83
  Post-Vaccination: A/H1N1: number analyzed (Participants) | 99 | 98 | 99 | 99
  Post-Vaccination: A/H1N1 | 93 | 98 | 99 | 99
  Post-Vaccination: A/H3N2 | 96 | 98 | 99 | 96
  Post-Vaccination: B Victoria | 88 | 98 | 98 | 99
  Post-Vaccination: B Yamagata: number analyzed (Participants) | 99 | 98 | 99 | 98
  Post-Vaccination: B Yamagata | 93 | 98 | 98 | 97

3. Primary Outcome: Number of Participants With Seroconversion or Significant Increase to Influenza Vaccine Antigens
Description: Anti-influenza antibodies were measured using HAI assay for 4 strains: H1N1, H3N2, B Victoria and B Yamagata. Seroconversion was defined as pre-vaccination titer <10 (1/dil) and post-vaccination titer >=40 (1/dil), and Significant increase was defined as pre-vaccination titer >=10 (1/dil) and >= 4-fold increase of post-vaccination titer.
Time Frame: 28 days post-final vaccination (post-vaccination)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years
Number analyzed (Participants) | 99 | 98 | 99 | 100
Participants
  A/H1N1: number analyzed (Participants) | 99 | 98 | 99 | 98
  A/H1N1 | 86 | 87 | 84 | 90
  A/H3N2 | 85 | 77 | 71 | 90
  B Victoria: number analyzed (Participants) | 99 | 97 | 99 | 98
  B Victoria | 84 | 87 | 95 | 92
  B Yamagata: number analyzed (Participants) | 99 | 98 | 99 | 97
  B Yamagata | 91 | 91 | 86 | 86

4. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions After Vaccination With Influenza Vaccine
Description: 1. Solicited injection site reactions:
     * Age 6-23 months: Tenderness, Erythema and Swelling(Grade 3: Tenderness: cries when injected limb is moved; Erythema and Swelling:>=50 mm)
     * Age >=2 years: Pain, Erythema and Swelling (Grade 3: Pain:unable to perform usual activities [age 2-11 years], significant interference with daily activities [age >=12 years]; Erythema and Swelling >=50 mm [age 2-11 years], >100 mm [age >=12 years])
  2. Solicited systemic reactions:
     * Age 6-23 months: Fever, Vomiting, Crying abnormal, Drowsiness, Appetite loss, Irritability (Grade 3: Fever:>39.5 degree Celsius; Vomiting:>=6 episodes/24 hours; Crying abnormal:>3 hours; Drowsiness:sleeping most of the time or difficult to wake up; Appetite loss: refuses >=3 feeds/meals or most feeds/meals; Irritability: inconsolable)
     * Age >=2 years:Fever, Headache, Malaise, Myalgia and Shivering (Grade 3:Fever>=39.0 degree Celsius; Headache, Malaise, Myalgia and Shivering:significant interference in daily activities)
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed using Safety Analysis Set which included all participants who received at least 1 dose of study vaccine. Here, 'Number Analyzed' = those participants with available data for specified categories. 'Number analyzed' = 0 signifies that reported reaction was not analyzed in the specified age group.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years
Number analyzed (Participants) | 100 | 100 | 100 | 100
Participants
  Injection site Pain / Tenderness | 12 | 40 | 35 | 24
  Grade 3: Injection site Pain / Tenderness | 0 | 0 | 0 | 0
  Injection site Erythema | 1 | 3 | 4 | 0
  Grade 3 Injection site Erythema | 0 | 0 | 0 | 0
  Injection site Swelling | 2 | 3 | 4 | 0
  Grade 3 Injection site Swelling | 0 | 0 | 0 | 0
  Fever: number analyzed (Participants) | 100 | 98 | 99 | 100
  Fever | 9 | 8 | 2 | 0
  Grade 3 Fever: number analyzed (Participants) | 100 | 98 | 99 | 100
  Grade 3 Fever | 0 | 2 | 0 | 0
  Vomiting: number analyzed (Participants) | 71 | 0 | 0 | 0
  Vomiting | 2 |  |  |
  Grade 3 Vomiting: number analyzed (Participants) | 71 | 0 | 0 | 0
  Grade 3 Vomiting | 2 |  |  |
  Crying abnormal: number analyzed (Participants) | 71 | 0 | 0 | 0
  Crying abnormal | 1 |  |  |
  Grade 3 Crying abnormal: number analyzed (Participants) | 71 | 0 | 0 | 0
  Grade 3 Crying abnormal | 0 |  |  |
  Drowsiness: number analyzed (Participants) | 71 | 0 | 0 | 0
  Drowsiness | 1 |  |  |
  Grade 3 Drowsiness: number analyzed (Participants) | 71 | 0 | 0 | 0
  Grade 3 Drowsiness | 0 |  |  |
  Appetite lost: number analyzed (Participants) | 71 | 0 | 0 | 0
  Appetite lost | 3 |  |  |
  Grade 3 Appetite lost: number analyzed (Participants) | 71 | 0 | 0 | 0
  Grade 3 Appetite lost | 0 |  |  |
  Irritability: number analyzed (Participants) | 71 | 0 | 0 | 0
  Irritability | 5 |  |  |
  Grade 3 Irritability: number analyzed (Participants) | 71 | 0 | 0 | 0
  Grade 3 Irritability | 0 | 0 |  |
  Headache: number analyzed (Participants) | 29 | 100 | 100 | 100
  Headache | 0 | 4 | 6 | 1
  Grade 3 Headache: number analyzed (Participants) | 29 | 100 | 100 | 100
  Grade 3 Headache | 0 | 1 | 0 | 0
  Malaise: number analyzed (Participants) | 29 | 100 | 100 | 100
  Malaise | 0 | 4 | 7 | 1
  Grade 3 Malaise: number analyzed (Participants) | 29 | 100 | 100 | 100
  Grade 3 Malaise | 0 | 0 | 0 | 0
  Myalgia: number analyzed (Participants) | 29 | 100 | 100 | 100
  Myalgia | 1 | 9 | 16 | 3
  Grade 3 Myalgia: number analyzed (Participants) | 29 | 100 | 100 | 100
  Grade 3 Myalgia | 0 | 0 | 0 | 0
  Shivering: number analyzed (Participants) | 29 | 100 | 100 | 100
  Shivering | 0 | 2 | 0 | 1
  Grade 3 Shivering: number analyzed (Participants) | 29 | 100 | 100 | 100
  Grade 3 Shivering | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) data were collected from Day 0 (post-vaccination) up to 28 days after the final vaccination (up to Day 56 for Group 1 and 2; Day 28 for Group 3 and 4)
Description: A solicited reaction is an AE that is prelisted in the electronic case report form (eCRF) and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and time to onset) prelisted (i.e., solicited) in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years | Quadrivalent Influenza Vaccine Group 4: >=18 Years
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 29/100 | 50/100 | 44/100 | 24/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quadrivalent Influenza Vaccine Group 1: 6 to 35 Months (N=100) | Quadrivalent Influenza Vaccine Group 2: 3 to 8 Years (N=100) | Quadrivalent Influenza Vaccine Group 3: 9 to 17 Years (N=100) | Quadrivalent Influenza Vaccine Group 4: >=18 Years (N=100)
Injection site pain (General disorders) | 12 | 40 | 35 | 24
Malaise (General disorders) | 0 | 4 | 7 | 1
Pyrexia (General disorders) | 14 | 8 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 9 | 16 | 3
Headache (Nervous system disorders) | 0 | 4 | 6 | 1
Irritability (Psychiatric disorders) | 6 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02451358/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02451358/SAP_001.pdf